CLINICAL TRIAL: NCT01314326
Title: Advanced Imaging for Glaucoma Study
Acronym: AIGS
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, David Huang, MD, PhD, Weeks Professor of Ophthalmic Research, Oregon Health & Science University, Oregon Health and Science University
Other Study IDs: OHSU IRB #00006611 - AIGS; R01EY013516 (NIH)
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma
Keywords: Optical Coherence Tomography; Glaucoma; Advanced Imaging
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Perimetric Glaucoma (PG): Patients with clinically confirmed abnormal VF and glaucomatous ONH or NFL defect
- Glaucoma Suspects and Pre-Perimetric Glaucoma (GSPPG) Group: Patients who are at high risk to develop perimetric glaucoma
- Normal Group: Volunteers with healthy eyes

SUMMARY:
The specific aims of the clinical studies are to:

1. Predict the development of glaucomatous visual field (VF) abnormality in glaucoma suspects and pre-perimetric glaucoma patients based on anatomic abnormalities detected by advanced imaging.
2. Predict the development of glaucomatous VF abnormality in glaucoma suspects and pre-perimetric glaucoma patients based on anatomic changes detected between successive advanced imaging tests.
3. Determine the sensitivity and specificity of glaucoma diagnosis based on advanced imaging tests.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of blindness in the US. Traditional methods of glaucoma diagnosis and monitoring lack good sensitivity and specificity. Delays in detecting glaucoma progression can lead to inadequate treatment and irreversible visual loss. Our goal is to improve glaucoma diagnosis by utilizing new imaging modalities that can reveal changes in the retinal layers affected by glaucoma and the associated reduction in retinal blood flow. Glaucoma selectively damages the retinal nerve fibers, which originate from cell bodies in ganglion cell layer (GCL) and travel to the optic nerve via the nerve fiber layer (NFL). We hypothesize that subtle damages in these structures can be detected earlier by optical coherence tomography (OCT) and other advanced imaging modalities than with current standard methods. OCT is based on infrared light reflectometry. It provides micrometer-scale cross-sectional images of retinal structures, which are not possible with other non-invasive techniques. More than 7,000 OCT systems are already being used for the diagnosis of glaucoma and retinal diseases. Phase I of the Advanced Imaging for Glaucoma (AIG) study demonstrated that peripapillary NFL thickness measured with the standard timedomain (TD) OCT technology has higher glaucoma diagnostic accuracy than other quantitative diagnostic technologies such as scanning laser polarimetry (SLP) and scanning laser tomography (SLT). We also demonstrated that more advanced diagnostic software and faster Fourier-domain (FD) OCT systems can achieve even better diagnostic accuracy and reproducibility. In the proposed Phase II of the AIG study, we will continue the most promising aspects of the research to further improve both technology and clinical practice.

The AIG Partnership investigators at the Oregon Health & Science University (OHSU), Massachusetts Institute of Technology (MIT), and University of Pittsburgh (UP) include those who invented OCT and pioneered its applications to glaucoma. OHSU, University of Southern California (USC), UP and University of Miami (UM) also have major glaucoma referral centers.

The Partnership combines engineers and clinicians who have the track record and synergy to develop novel technologies, evaluate them in a rigorous clinical study, and transfer the knowledge to industry and medicine.

The Specific Aims of this competing renewal proposal are:

1. Develop image processing and diagnostic analysis for 3-dimensional OCT data. The AIG study is currently using 26 kHz (axial scan repetition rate) FD-OCT technology that is capable of scanning the macula and the optic nerve head in a fraction of a second. We have completed computer algorithms for mapping and analysis of the macular ganglion cell complex (mGCC) and the peripapillary NFL, which lead to significant improvement in diagnostic accuracy. We propose to continue the work on disc cupping analysis, NFL reflectivity analysis, and expert system combination of multiple anatomic parameters to further improve diagnostic accuracy. Algorithms to detect progression of glaucoma over time are also planned.
2. Develop ultrafast OCT systems for imaging of the macula and optic nerve head. Although current FD-OCT technology at 26 kHz represents a tremendous advance over standard 400 Hz TD-OCT (Zeiss Stratus), it still takes ~4 seconds for a full 3-dimensional (3D) raster scan of the macula. Our goal is to reduce this time to 0.1-0.2 second so 3D scans will be minimally affected by eye movement. This requires an ultrafast speed of 500-1000 kHz. We plan to adapt the Fourier-domain modelocked-laser (FDML) swept-source OCT, which has already been demonstrated at 249 kHz at MIT. We will further improve its speed to 500 kHz. The short integration time and phase stability of FDML-OCT is ideal for Doppler perfusion measurement (see next aim). For an even faster speed, parallel line-scan FD-OCT at 1 MHz will be developed. Line-scan OCT is not suitable for Doppler flow measurement due to the relatively long integration time, but is more efficient for ultrafast anatomic imaging. It will allow full 8x8 mm macular 3D imaging in 0.2 second. We will also continue to develop polarization-sensitive (PS) OCT for NFL birefringence measurement, which will also be greatly enhanced by higher speed and greater averaging to suppress noise.
3. Develop Doppler OCT to measure retinal perfusion. One of the significant achievements of the AIG project is the demonstration of a reproducible method of measuring total retinal blood flow using Doppler FD-OCT. Reduced flow was found in glaucomatous eyes, opening an important new approach to measure the severity of glaucoma and assess the risk for further progression. An automated algorithm will be developed to improve the robustness of Doppler flow measurement. We will also investigate Doppler OCT with the ultrafast FDML-OCT system.
4. Evaluate OCT technologies in a longitudinal clinical study. An extension of the ongoing clinical study is proposed. Participants (1000 planned with 700+ already enrolled) in normal, glaucoma suspect, and glaucoma groups will be followed. OCT and other imaging technologies will be compared for diagnostic accuracy, detection of early progression, and prediction of future visual field loss. The impact of intraocular pressure on retinal blood flow and how flow affects the risk of glaucoma will also be studied.

Quantitative imaging technologies such as OCT have improved glaucoma management by reducing reliance on insensitive tests such as perimetry and subjective disc grading. The AIG Partnership comprises engineers and clinicians who co-invented OCT. We propose to further improve its performance with higher speed, more sophisticated software, and novel functional measurements. The eventual goal is to save vision by basing glaucoma treatment decisions on speedy and reliable imaging tests.

ELIGIBILITY:
Inclusion Criteria for Normal Participants:

* No history of glaucoma, retinal pathology, keratorefractive surgery, or corticosteroid use.
* Normal visual field (VF), intraocular pressure (IOP), optic nerve head and nerve fiber layer.
* Central pachymetry > 500 μm.
* Open angle.

Inclusion Criteria for Glaucoma Suspects & Pre-Perimetric Glaucoma Participants:

* Ocular hypertension, defined as IOP ≥ 24 mmHg in one eye and IOP ≥ 22 mmHg in the fellow eye, on or off glaucoma medications.
* Optic nerve head (ONH) or nerve fiber layer (NFL) defect visible on slit-lamp biomicroscopy and stereo color fundus photography as defined for the PG group.
* The fellow eye meeting the eligibility criteria for the PG group.
* GSPPG eyes must not have an abnormal VF as defined for the PG group.
* GSPPG participants having glaucomatous ONH or NFL defect are subclassified as PPG; the remainder are subclassified as GS.

Inclusion Criteria for Perimetric Glaucoma Participants:

* Abnormal VF and
* Glaucomatous ONH of NFL defect.

Exclusion Criteria Common to All Groups:

* Best corrected visual acuity worse than 20/40.
* Age < 40 or > 79 years.
* Refractive error > +3.0D or < -7.0 D.
* Previous intraocular surgery except for uncomplicated cataract extraction with posterior chamber IOL implantation.
* Diabetic retinopathy or other disease that may cause visual field loss or optic disc abnormalities.
* Inability to clinically view or photograph the optic discs due to media opacity or poorly dilating pupil.
* Inability to obtain advanced imaging data with acceptable quality or reliable VF test results.
* Life-threatening or debilitating illness making it unlikely patient could successfully complete the study.
* Refusal of informed consent or of commitment to the full length of the study.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll both males and females and include all ethnic and racial groups through clinical practices in the centers. The study will enroll subjects in the older adult age range commonly affected by glaucoma - 40 years or older. The study will exclude people with life-threatening or debilitating illness that would make 5-year participation unlikely or cooperation with tests difficult. For similar reasons those older than 79 years are excluded. The study also excludes those with any disease that might confound the diagnosis of glaucoma. Otherwise people with any health status are eligible for enrollment. Three groups of participants are recruited in the AIG study: normal (N), glaucoma suspects & preperimetric glaucoma (GSPPG) and perimetric glaucoma (PG).
Sampling Method: Non-Probability Sample
Enrollment: 832 (Actual)
Dates: Start 2003-09; Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

PRIMARY OUTCOMES:
Developing glaucoma or progression with glaucoma as defined by study criteria | 5 years or the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Study Chair — Oregon Health and Science University; Joel S. Schuman, MD, Principal Investigator — University of Pittsburgh; Rohit Varma, MD, Principal Investigator — University of Southern California; David S. Greenfield, MD, Principal Investigator — University of Miami; John Morrison, MD, Principal Investigator — Oregon Health and Science University; James Fujimoto, PhD, Principal Investigator — Massachusettes Inistitute of Technology
Locations (5):
- United States (5):
  - University of Southern California, Doheny Eye Institute, Los Angeles, California
  - University of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - Massachusettes Institute of Technology, Boston, Massachusetts
  - Oregon Health & Science University, Casey Eye Institute, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Tan O, Li G, Lu AT, Varma R, Huang D; Advanced Imaging for Glaucoma Study Group. Mapping of macular substructures with optical coherence tomography for glaucoma diagnosis. Ophthalmology. 2008 Jun;115(6):949-56. doi: 10.1016/j.ophtha.2007.08.011. Epub 2007 Nov 5. PMID 17981334
- [Background] Potsaid B, Baumann B, Huang D, Barry S, Cable AE, Schuman JS, Duker JS, Fujimoto JG. Ultrahigh speed 1050nm swept source/Fourier domain OCT retinal and anterior segment imaging at 100,000 to 400,000 axial scans per second. Opt Express. 2010 Sep 13;18(19):20029-48. doi: 10.1364/OE.18.020029. PMID 20940894
- [Background] Grzywacz NM, de Juan J, Ferrone C, Giannini D, Huang D, Koch G, Russo V, Tan O, Bruni C. Statistics of optical coherence tomography data from human retina. IEEE Trans Med Imaging. 2010 Jun;29(6):1224-37. doi: 10.1109/TMI.2009.2038375. Epub 2010 Mar 18. PMID 20304733
- [Background] Tan O, Chopra V, Lu AT, Schuman JS, Ishikawa H, Wollstein G, Varma R, Huang D. Detection of macular ganglion cell loss in glaucoma by Fourier-domain optical coherence tomography. Ophthalmology. 2009 Dec;116(12):2305-14.e1-2. doi: 10.1016/j.ophtha.2009.05.025. Epub 2009 Sep 10. PMID 19744726
- [Background] Sung KR, Wollstein G, Schuman JS, Bilonick RA, Ishikawa H, Townsend KA, Kagemann L, Gabriele ML; Advanced Imaging in Glaucoma Study Group. Scan quality effect on glaucoma discrimination by glaucoma imaging devices. Br J Ophthalmol. 2009 Dec;93(12):1580-4. doi: 10.1136/bjo.2008.152223. Epub 2009 Aug 18. PMID 19692363
- [Background] Wang Y, Lu A, Gil-Flamer J, Tan O, Izatt JA, Huang D. Measurement of total blood flow in the normal human retina using Doppler Fourier-domain optical coherence tomography. Br J Ophthalmol. 2009 May;93(5):634-7. doi: 10.1136/bjo.2008.150276. Epub 2009 Jan 23. PMID 19168468
- [Background] Wang Y, Fawzi AA, Varma R, Sadun AA, Zhang X, Tan O, Izatt JA, Huang D. Pilot study of optical coherence tomography measurement of retinal blood flow in retinal and optic nerve diseases. Invest Ophthalmol Vis Sci. 2011 Feb 11;52(2):840-5. doi: 10.1167/iovs.10-5985. Print 2011 Feb. PMID 21051715
- [Background] Zhao M, Izatt JA. Single-camera sequential-scan-based polarization-sensitive SDOCT for retinal imaging. Opt Lett. 2009 Jan 15;34(2):205-7. doi: 10.1364/ol.34.000205. PMID 19148256
- [Background] Greenfield DS, Weinreb RN. Role of optic nerve imaging in glaucoma clinical practice and clinical trials. Am J Ophthalmol. 2008 Apr;145(4):598-603. doi: 10.1016/j.ajo.2007.12.018. Epub 2008 Mar 4. PMID 18295183
- [Background] Mumcuoglu T, Townsend KA, Wollstein G, Ishikawa H, Bilonick RA, Sung KR, Kagemann L, Schuman JS Manuscript #AJO-08-106. Am J Ophthalmol Accepted for Publication: May 28, 2008.
- [Background] Alasil T, Tan O, Lu AT, Huang D, Sadun AA. Correlation of Fourier domain optical coherence tomography retinal nerve fiber layer maps with visual fields in nonarteritic ischemic optic neuropathy. Ophthalmic Surg Lasers Imaging. 2008 Jul-Aug;39(4 Suppl):S71-9. doi: 10.3928/15428877-20080715-03. PMID 18777877
- [Background] Asrani S, Sarunic M, Santiago C, Izatt J. Detailed visualization of the anterior segment using fourier-domain optical coherence tomography. Arch Ophthalmol. 2008 Jun;126(6):765-71. doi: 10.1001/archopht.126.6.765. PMID 18541838
- [Background] Memarzadeh F, Tang M, Li Y, Chopra V, Francis BA, Huang D. Optical coherence tomography assessment of angle anatomy changes after cataract surgery. Am J Ophthalmol. 2007 Sep;144(3):464-5. doi: 10.1016/j.ajo.2007.04.009. PMID 17765435
- [Background] Wang Y, Bower BA, Izatt JA, Tan O, Huang D. In vivo total retinal blood flow measurement by Fourier domain Doppler optical coherence tomography. J Biomed Opt. 2007 Jul-Aug;12(4):041215. doi: 10.1117/1.2772871. PMID 17867804
- [Background] Sehi M, Ume S, Greenfield DS. Scanning laser polarimetry with enhanced corneal compensation and optical coherence tomography in normal and glaucomatous eyes. Invest Ophthalmol Vis Sci. 2007 May;48(5):2099-104. doi: 10.1167/iovs.06-1087. PMID 17460267
- [Background] Pedersen CJ, Huang D, Shure MA, Rollins AM. Measurement of absolute flow velocity vector using dual-angle, delay-encoded Doppler optical coherence tomography. Opt Lett. 2007 Mar 1;32(5):506-8. doi: 10.1364/ol.32.000506. PMID 17392903
- [Background] Memarzadeh F, Li Y, Chopra V, Varma R, Francis BA, Huang D. Anterior segment optical coherence tomography for imaging the anterior chamber after laser peripheral iridotomy. Am J Ophthalmol. 2007 May;143(5):877-9. doi: 10.1016/j.ajo.2006.11.055. Epub 2006 Dec 29. PMID 17452177
- [Background] Sadda SR, Tan O, Walsh AC, Schuman JS, Varma R, Huang D. Automated detection of clinically significant macular edema by grid scanning optical coherence tomography. Ophthalmology. 2006 Jul;113(7):1187.e1-12. doi: 10.1016/j.ophtha.2005.12.020. Epub 2006 May 2. PMID 16647123
- [Background] Huang XR, Knighton RW, Shestopalov V. Quantifying retinal nerve fiber layer thickness in whole-mounted retina. Exp Eye Res. 2006 Nov;83(5):1096-101. doi: 10.1016/j.exer.2006.05.020. Epub 2006 Jul 7. PMID 16828473
- [Background] Sarunic MV, Applegate BE, Izatt JA. Real-time quadrature projection complex conjugate resolved Fourier domain optical coherence tomography. Opt Lett. 2006 Aug 15;31(16):2426-8. doi: 10.1364/ol.31.002426. PMID 16880844
- [Background] Sehi M, Greenfield DS. Assessment of retinal nerve fiber layer using optical coherence tomography and scanning laser polarimetry in progressive glaucomatous optic neuropathy. Am J Ophthalmol. 2006 Dec;142(6):1056-9. doi: 10.1016/j.ajo.2006.07.043. Epub 2006 Sep 5. PMID 17157591
- [Background] Huang XR, Knighton RW. Microtubules contribute to the birefringence of the retinal nerve fiber layer. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4588-93. doi: 10.1167/iovs.05-0532. PMID 16303953
- [Derived] Loewen NA, Zhang X, Tan O, Francis BA, Greenfield DS, Schuman JS, Varma R, Huang D; Advanced Imaging for Glaucoma Study Group. Combining measurements from three anatomical areas for glaucoma diagnosis using Fourier-domain optical coherence tomography. Br J Ophthalmol. 2015 Sep;99(9):1224-9. doi: 10.1136/bjophthalmol-2014-305907. Epub 2015 Mar 20. PMID 25795917
- [Derived] Sehi M, Goharian I, Konduru R, Tan O, Srinivas S, Sadda SR, Francis BA, Huang D, Greenfield DS. Retinal blood flow in glaucomatous eyes with single-hemifield damage. Ophthalmology. 2014 Mar;121(3):750-8. doi: 10.1016/j.ophtha.2013.10.022. Epub 2013 Nov 28. PMID 24290800
- [Derived] Sehi M, Zhang X, Greenfield DS, Chung Y, Wollstein G, Francis BA, Schuman JS, Varma R, Huang D; Advanced Imaging for Glaucoma Study Group. Retinal nerve fiber layer atrophy is associated with visual field loss over time in glaucoma suspect and glaucomatous eyes. Am J Ophthalmol. 2013 Jan;155(1):73-82.e1. doi: 10.1016/j.ajo.2012.07.005. Epub 2012 Oct 1. PMID 23036570
- See also: AIGS main website — http://www.aigstudy.net/